## Statistical Analysis Plan (SAP)

## Section 1: Administrative

| Section/Item | Index | Description |
|---|---|---|
| Title and trial registration | 1a | Assessment of prospective CYP2C19 genotype guided<br><u>Dosing of Anti-Platelet Therapy in Percutaneous Coronary</u> |
| | 1b | Intervention (ADAPT) Clinical trials.gov registration: NCT02508116 |
| CAD Version | 2 | CAD Version 4.0 December 2017 |
| SAP Version | 2 | SAP Version 1.0 December 2017 |
| Protocol version | 3. | Protocol Version 3.0 date June 1, 2017 |
| SAP revisions | 4 | No prior changes were made to the SAP. SAP was drafted after study completion. |
| SAP contributors | 5 | Sony Tuteja, PharmD, Co-Pl<br>Jay Giri, MD, Co-Pl<br>Henry Glick, PhD, Biostatistician |
| Signatures | 6 | Sony Tuteja |
| | | Jay Giri |
| | | Henry Glick |

Section 2: Introduction

| Section/Item | Index | Description |
|---|---|---|
| Background and Introduction | 7 | Clopidogrel is a thienopyridine antiplatelet agent, which inhibits the purinergic P2Y12 receptor on platelets and prevents their aggregation. It is commonly used in patients with acute coronary syndromes (ACS) undergoing percutaneous coronary intervention (PCI). <i>CYP2C19</i> is one of the principal enzymes involved in the bioactivation of clopidogrel from the pro-drug to its active metabolite. The most common loss of function (LOF) allele is *2 (c.681G>A; rs4244285), with frequencies of ~15% in Caucasians and Africans and 29-35% in Asians. A large meta-analysis performed by Mega and colleagues demonstrated that CYP2C19*2 carriers treated with clopidogrel have a higher risk for major adverse cardiac events compared to noncarriers (hazard ratio (HR) of 1.55, 95%CI 1.11-2.17 for heterozygotes; HR 1.76, 95% CI 1.24-2.50) and higher risk of stent thrombosis (HR 2.67, 95% CI 1.69-4.22 for heterozygotes; HR 3.97, 95% CI 1.75-9.02 for homozygotes). Therefore, clopidogrel is less effective in patients who are CYP2C19 poor metabolizers and alternative therapy is recommended. While a body of observational literature and clinical guidelines² suggest prescribing alternative antiplatelet therapy in carriers of <i>CYP2C19</i> LOF alleles, it is unknown whether physicians will follow genotype guided recommendations when pharmacogenetic (PGx) results are presented to them in a real world setting. To provide evidence regarding the implementation and effectiveness of PGx testing following PCI, we examined the differences in prescribing of antiplatelet drugs when presented with genotype data. We also evaluated physician's adherence to the genotype guided antiplatelet recommendations. |
| Objectives | 8 | <ol> <li>To determine the effect of CYP2C19 genotyping on the prescribing patterns of antiplatelet therapies following cardiac catheterization.</li> <li>To determine the rates of clinical outcomes.</li> <li>To identify factors linked with successful implementation of clinical pharmacogenetic (PGx) testing in a large academic medical center.</li> </ol> |

Section 3: Study Methods

| Section/Item | Index | Description |
|---|---|---|
| Trial Design | 9 | This was a prospective, pragmatic, randomized, controlled clinical pharmacogenetic implementation trial. Patients undergoing PCI with stent implantation requiring anti-platelet therapy were randomized 1:1 to either rapid genotyping of <i>CYP2C19</i> with reporting of results to the interventional cardiologist or no genotyping (usual care). |
| Randomization | 10 | We used Stata's V13.1 (College Lake, TX) random number generator to draw random numbers that were used to randomize participants to the genotyping and usual care groups. Randomization was stratified by hospital site and by the presence or absence of ACS. Acute coronary syndrome was defined as unstable angina, non-ST elevation myocardial infarction, or ST-elevation myocardial infarction. The designation of ACS vs. stable angina was made by the treating interventional cardiologist. Within each of the four groups, randomization was balanced so that after every 10 patients, 5 were randomized to the genotyped group and 5 to usual care. |
| Sample size | 11 | The sample size calculation was based on two factors: 1) the rate of pre-study prasugrel/ticagrelor use (20%) and 2) anticipated increase in prasugrel/ticagrelor prescribing based on the frequency <i>CYP2C19</i> LOF variants (~30-35%). We estimated a 15% difference in the use of prasugrel/ticagrelor in the two groups (35% in the genotyped group and 20% in the control group). A sample size of 138 per group (a total of 276) would provide 80% power at an alpha level of 0.05 to detect this difference. We increased our sample size to ~250 per group to allow for subgroup comparisons (e.g. ACS vs. stable coronary disease). |
| Framework | 12 | Genotyping will increase the prescribing of prasugrel or ticagrelor from the baseline rate of 20%. |
| Statistical interim analyses and stopping guidance | 13 | No interim analyses planned. |
| Timing of final analysis | 14 | Participants were followed until May 31, 2017 for prospective clinical endpoints assessment with the intention of a 12 month follow-up time for each participant. All analyses were performed collectively after May 31, 2017. |
| Timing of outcome assessment | 15 | Participants were called by telephone every 3 months ± 2 weeks following randomization to assess occurrence of clinical endpoints. Medical records were requested for admissions that occurred outside UPHS. Medical records within UPHS were reviewed simultaneously to assess additional clinical outcomes not reported by participants. |

Section 4: Statistical Principles

| Section/Item | Index | Description |
|---|---|---|
| Confidence | 16 | The primary outcome was claimed at an alpha level of p=0.05. |
| intervals and p- | 17 | No corrections were made for multiple testing. |
| value | 18 | Confidence intervals pertaining to the probability of receipt of |
| | | antiplatelet agents were reported. |
| Adherence and | 19a | Adherence to the genotype guided recommendations was |
| protocol deviations | | assessed in the genotyped group by comparing the discharge |
| | | antiplatelet medication to those recommended by the CPIC |
| | | guidelines. The research coordinator asked the prescribing |
| | | cardiologists to provide any reasons for non-adherence. |
| | | Adherence was not described in the usual care group as |
| | | prescribing decisions were made by the cardiologist as per usual |
| | | care. |
| | 19b | The adherence rate was defined as the number of participants in |
| | | genotyped group with LOF variants that received prasugrel or |
| | | ticagrelor + the number of participants without these variants that |
| | 4.0 | received clopidogrel divided by the total number in this group |
| | 19c | The only protocol deviations that were encountered in this trial |
| | | were enrollment of participants that did not meet the |
| | | inclusion/exclusion criteria. Since this was a pragmatic clinical |
| | | trial, most of the procedures were performed within the context of usual care. |
| | 104 | |
| | 19d | Participants that did not meet inclusion/exclusion criteria and |
| | | were withdrawn from the study by the treating physician or study staff. |
| Analysis | 20 | |
| Analysis | 20 | Modified intent to treat (removing the participants that did not |
| population | | meet the inclusion criteria). |

Section 5: Trial Population

| Section/Item | Index | Description |
|---|---|---|
| Screening data | 21 | The number of PCIs performed, participants screened, and |
| | | reasons for screening failure were collected by each study site. |
| | | These data were reviewed by study staff to monitor recruitment |
| | | and enrollment progress throughout the study. |
| Eligibility | 22 | Inclusion Criteria |
| | | 1. Male and female subjects, ≥18 to ≤80 years at time of study |
| | | Status post PCI with stent implantation requiring antiplatelet therapy |
| | | 3. Willingness to comply with all study-related procedures |
| | | Exclusion criteria: |
| | | <ol> <li>Pending imminent surgery placing patients at increased risk<br/>for bleeding with prasugrel or ticagrelor.</li> </ol> |
| | | 2. History of intracranial hemorrhage, TIA, and stroke |
| | | 3. Active bleeding |
| | | 4. Need for long-term anticoagulation (i.e. warfarin, |
| | | dabigatran, rivaroxaban, apixaban, edoxaban, or lovenox). |
| | | 5. Current or prior (within the past four weeks) treatment with |
| | | voraxapar (Zontivity). |
| | | Severe renal or hepatic impairment |
| | | 7. Treating physician does not want subject to participate |
| Recruitment | 23 | The number of participants assessed for eligibility along with reasons for non-enrollment will be reported as available. |
| Withdrawal/ follow-<br>up | 24a | The numbers of withdrawal from follow-up clinical assessments were reported as the intervention is a one-time event. |
| αp | 24b | The number and time post randomization of voluntary |
| | 210 | withdrawals by participants or lost to follow-up were reported. |
| | 24c | Reasons for voluntary withdrawal or lost to follow-up were |
| | | reported if available. |
| Baseline patient | 25a | Sex, race, age, hospital site, presence of acute coronary |
| characteristics | | syndrome (ACS), insurance type, work status, tobacco use, past |
| | | medical history, medications prior to admission. |
| | 25b | For categorical variables, frequencies and percentages were |
| | | reported. For continuous variables, the number of subjects, mean |
| | | and standard deviation were reported by randomization group. |

Section 6: Analysis

| Section/Item | Index | Description |
|---|---|---|
| Outcome | 26a | Primary outcome: |
| definitions | | The number and proportion of participants receiving |
| | | prasugrel/ticagrelor at discharge from index PCI in each randomized. |
| | | Timing <7 days |
| | | Timing a days |
| | | Secondary Outcomes: |
| | | Adherence to the CPIC guideline suggested antiplatelet |
| | | therapy recommendations based on genotype (intervention |
| | | group only). Timing <7 days. |
| | | Major adverse cardiac events (MACE) defined as |
| | | cardiovascular death, myocardial infarction, stroke, urgent |
| | | need for revascularization, and stent thrombosis (Academic |
| | | Research Consortium "definite" stent thrombosis (** teddermo |
| | | last follow-up. |
| | | Major bleeding events as defined by the Bleeding Academic |
| | | Research Consortium (BARC) <sup>4</sup> type 3 or 5. Timing at last |
| | | follow-up. |
| | | 4. Non-cardiac mortality. Timing at last follow-up. |
| | | 5. Implementation Metrics. Timing at last follow-up. |
| | | a. Genotype test turnaround time (Time result reported |
| | | to physician – time of buccal swab). |
| | | b. Number of inconclusive results. |
| | 26h | |
| | 26b<br>26c | n/a Time to MACE or major bleed |
| Analysis methods | 27a | Primary outcome: |
| Analysis memous | 21a | Discharge antiplatelet therapy choice by genotyped and usual care |
| | | group was compared using the chi-square or Fisher's exact test. The |
| | | probability of receipt of antiplatelet agents was determined by logistic |
| | | regression. |
| | | regression. |
| | | Secondary outcomes: |
| | | The adherence rate to the genotype guided recommendations |
| | | for the genotyped group was determined by reporting the number |
| | | of participants with LOF variants that received prasugrel or |
| | | ticagrelor + the number of participants without these variants that |
| | | received clopidogrel divided by the total number in the genotyped |
| | | arm. |
| | | 2. Clinical outcomes. Frequencies of CV related death, MI, stroke |
| | | urgent, need for revascularization and stent thrombosis was |
| | | reported as well frequencies of bleeding complications and |
| | | compared using chi-square test or Fisher's exact test when |
| | | appropriate. The time to first major cardiac event as a composite |
| | | endpoint (CV related death, MI, stroke urgent need for |
| | | revascularization and stent thrombosis) was determined. The |
| | | incidence of first MACE and first major bleeding events between |
| | | the groups was compared by use of Kapan-Meier estimators and |
| | | statistical tests evaluated based on log-rank tests. |
| | | 3. Implementation. The turnaround time for test result in the |
| | <u> </u> | o. Implementation. The turnaround time for test result in the |

| | | genotyped group was presented as mean ± standard deviation |
|---|---|---|
| | | (hours). |
| | 27b | n/a |
| | 27c | n/a |
| | 27d | n/a |
| | 27e | n/a |
| | 27f | To evaluate whether genotyping influenced MACE outcomes in participants with ACS, an interaction term between ACS and group assignment was tested in a Cox proportional hazard model. |
| Missing data | 28 | For time to MACE analysis, participants were censored at the date of event or time of known last follow-up. |
| Additional analyses | 29 | Post-hoc analyses Genotype was determined in the control group at the end of the trial. We combined the groups and evaluated outcomes by CYP2C19 genotype and antiplatelet drugs prescribed at discharge. Participants were grouped into the following categories: 1) Carriers of normal function alleles receiving any antiplatelet drug, 2) LOF carriers receiving clopidogrel, or 3) LOF carriers receiving prasugrel or ticagrelor. Time to MACE, major bleeding and a composite safety/efficacy endpoint consisting of MACE, major bleeding and non-cardiac mortality was determined in the three groups. Cox proportional hazards models were used to assess the effects of having an LOF allele and receiving clopidogrel therapy, having an LOF allele and receiving alternative therapy, and not having an LOF allele on the occurrence of first MACE, first major bleed, and first composite outcome. The Cox model was controlled for age at entry to the study, the date of catheterization, gender, race, hospital site, and history of ACS, smoking, hypertension, diabetes, and myocardial infarction. |
| Harms | 30 | No harms as a result of the genotyping intervention were reported. |
| Statistical software | 31 | Stata's V13.1 (College Lake, TX) |
| References | 32 | <ol> <li>Mega, J.L. et al. Reduced-function CYP2C19 genotype and risk of adverse clinical outcomes among patients treated with clopidogrel predominantly for PCI: a meta-analysis. JAMA 304, 1821-30 (2010).</li> <li>Scott, S.A. et al. Clinical Pharmacogenetics Implementation Consortium Guidelines for CYP2C19 Genotype and Clopidogrel Therapy: 2013 Update. Clin Pharmacol Ther 94, 317-23 (2013).</li> <li>Mauri, L., Hsieh, W.H., Massaro, J.M., Ho, K.K., D'Agostino, R. &amp; Cutlip, D.E. Stent thrombosis in randomized clinical trials of drug-eluting stents. N Engl J Med 356, 1020-9 (2007).</li> <li>Mehran, R. et al. Standardized Bleeding Definitions for Cardiovascular Clinical Trials: A Consensus Report From the Bleeding Academic Research Consortium. Circulation 123, 2736-47 (2011).</li> </ol> |